CLINICAL TRIAL: NCT01650779
Title: Evaluation of Glycosphingolipid Clearance in Patients Treated With Agalsidase Alfa Who Switch to Agalsidase Beta (The INFORM Study)
Brief Title: A Study Evaluating Glycosphingolipid Clearance in Patients Treated With Agalsidase Alfa Who Switch to Agalsidase Beta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGAL19412
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-06

CONDITIONS: Fabry Disease
Keywords: alpha-galactosidase A; a-GAL; Fabry; GL-3; Fabrazyme
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Agalsidase beta (Experimental)
  Interventions: Biological: Agalsidase beta

INTERVENTIONS:
Biological: Agalsidase beta — Commercially available agalsidase beta 1.0 mg/kg administered as an intravenous infusion q2w up to Month 6.
  Other Names: Fabrazyme®

SUMMARY:
This is an exploratory study to evaluate changes in glycosphingolipid levels and other (exploratory) Fabry disease parameters in male Fabry disease participants who were previously treated with agalsidase alfa (Replagal®) 0.2 milligram per kilogram (mg/kg) every two weeks (q2w) and who are being switched to agalsidase beta (Fabrazyme®) 1.0 mg/kg q2w.

ELIGIBILITY:
Inclusion Criteria:

* The participant and/or his parent/legal guardian is willing and able to provide signed informed consent, and the participant, if less than (<) 18 years of age, is willing to provide assent if deemed able to do so
* Participant is male and has been treated with agalsidase alfa at 0.2 mg/kg q2w for the 12 months prior to switching to agalsidase beta
* The participant has a confirmed diagnosis of Fabry disease by alfa-galactosidase A (alfa-GAL) activity and/or genotyping per local standards
* The participant when switched to agalsidase beta receives the labeled dose, that is, 0.9 to 1.1 mg/kg (1 mg/kg) q2w, and must be willing to maintain the labeled dose for the duration of the study

Exclusion Criteria:

* The participant is on dialysis or is post renal transplantation
* The participant is in end-stage cardiac failure
* The participant and/or his parent or legal guardian, in the opinion of the investigator, is unable to adhere to the requirements of the study
* The participant has been switched from agalsidase alfa to agalsidase beta and does not have historical blood and urine samples

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- United States (6):
  - Coral Springs, Florida
  - Decatur, Georgia
  - Baltimore, Maryland
  - Grand Rapids, Michigan
  - Hellertown, Pennsylvania
  - Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in the United States of America between April 30, 2012 and March 15, 2013.
Pre-assignment Details: A total of 16 participants were screened of which 1 participant was screen failure. A total of 15 participants were enrolled in this study.
Groups:
- Agalsidase Beta: Commercially available agalsidase beta (Fabrazyme ®) 1.0 milligram per kilogram (mg/kg) administered as an intravenous infusion every 2 weeks (q2w) up to Month 6.
Period: Overall Study
Arm/Group | Agalsidase Beta
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants were included in the analysis.
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (16.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 13
  Hispanic | 1
  Other | 1
Duration of Fabry Disease [Median (Full Range); unit: years] — Duration of Fabry disease was calculated from date of initial diagnosis of Fabry disease to date of the first study infusion. Number of participants analyzed for this baseline measure were 14, as one participant did not have information on date of initial diagnosis of Fabry disease.
  years | 9.3 (4.73) [2 to 19]
Method of Diagnosis of Fabry Disease [Number; unit: participants] — Number of participants with each method (genotype, leukocyte alfa-galactosidase A [GAL] activity, and plasma alfa-GAL activity) are reported. Some participants were diagnosed by more than 1 method, hence reported under more than 1 category.
  participants
    Genotype | 14
    Leukocyte alfa-galactosidase A (GAL) activity | 11
    Plasma alfa-GAL activity | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Plasma Deacylated Globotriaosylceramide (Lyso-GL-3) at Month 2, 4 and 6
Description: Percent change from baseline = ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. For levels reported as below quantitative limit (BQL), the lower limit of quantitation (LLOQ) value was divided by 2 and used in the calculation to estimate values in samples that were BQL. The LLOQ for plasma lyso-GL-3 was 5.0 nanogram per milliliter (ng/mL). This study is exploratory because little is known about the dose-response of these biomarkers to enzyme replacement therapy (ERT) or about the clinical significance of the biomarkers.
Time Frame: Baseline, Month 2, 4, 6
Population: All enrolled participants were included in the analysis. Here, 'n' signifies participants with plasma Lyso-GL-3 assessment at the specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 15
percent change
  Month 2 (n=14) | -31.71 (22.540)
  Month 4 (n=12) | -39.04 (22.280)
  Month 6 (n=14) | -39.54 (23.567)
Statistical Analysis 1: Comparison: Agalsidase Beta; Baseline versus Month 2: Analysis was performed using one sample t-test; Test type: Superiority or Other; p = 0.0002, One sample t-test
Statistical Analysis 2: Comparison: Agalsidase Beta; Baseline versus Month 4: Analysis was performed using one sample t-test; Test type: Superiority or Other; p < 0.0001, One sample t-test
Statistical Analysis 3: Comparison: Agalsidase Beta; Baseline versus Month 6: Analysis was performed using one sample t-test; Test type: Superiority or Other; p < 0.0001, One sample t-test

2. Secondary Outcome: Percent Change From Baseline in Plasma Globotriaosylceramide (GL-3) at Month 2, 4 and 6
Description: Percent change from baseline = ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. For levels reported as BQL, the LLOQ value was divided by 2 and used in the calculation to estimate values in samples that were BQL. The LLOQ for plasma GL-3 was 2.0 microgram per milliliter (mcg/mL). This study is exploratory because little is known about the dose-response of these biomarkers to ERT or about the clinical significance of the biomarkers.
Time Frame: Baseline, Month 2, 4, 6
Population: All enrolled participants were included in the analysis. Here, 'n' signifies participants with plasma GL-3 assessment at the specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 15
percent change
  Month 2 (n=12) | -10.33 (21.087)
  Month 4 (n=10) | -12.80 (23.388)
  Month 6 (n=12) | -17.89 (25.291)
Statistical Analysis 1: Comparison: Agalsidase Beta; Baseline versus Month 2: Analysis was performed using one sample t-test; Test type: Superiority or Other; p = 0.1178, One sample t-test
Statistical Analysis 2: Comparison: Agalsidase Beta; Baseline versus Month 4: Analysis was performed using one sample t-test; Test type: Superiority or Other; p = 0.1176, One sample t-test
Statistical Analysis 3: Comparison: Agalsidase Beta; Baseline versus Month 6: Analysis was performed using one sample t-test; Test type: Superiority or Other; p = 0.0322, One sample t-test

3. Secondary Outcome: Percent Change From Baseline in Urine GL-3 at Month 2, 4, and 6
Description: Percent change from baseline = ([post-baseline value minus baseline value] divided by [baseline value]) multiplied by 100. For levels reported as BQL, the LLOQ value was divided by 2 and used in the calculation to estimate values in samples that were BQL. The LLOQ for urine GL-3 was 0.2 mcg/mL. The absolute values were calculated in microgram per millimole (mcg/mmol) of creatinine by dividing GL-3 (mcg/mL) by creatinine (mg/mL) and multiplying by 113.13 (mg/mmol), the molecular weight of creatinine. For levels reported BQL, the absolute values were calculated in microgram per millimole (mcg/mmol) of creatinine by dividing 0.1 (mcg/mL) by creatinine (mg/mL) and multiplying by 133.13 (mg/mmol). This study is exploratory because little is known about the dose-response of these biomarkers to ERT or about the clinical significance of the biomarkers.
Time Frame: Baseline, Month 2, 4, 6
Population: All enrolled participants were included in the analysis. Here, 'n' signifies participants with urine GL-3 assessment at the specified time point.
Measure: Median (Full Range); unit: percent change
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 15
percent change
  Month 2 (n=13) | -44.71 [-98.4 to 1068.2]
  Month 4 (n=12) | -41.49 [-96.5 to 464.9]
  Month 6 (n=12) | -33.75 [-97.1 to 1116.7]
Statistical Analysis 1: Comparison: Agalsidase Beta; Baseline versus Month 2: Analysis was performed using one sample test of median (sign test). The percent change and absolute change from baseline in urine GL-3 levels were not normally distributed and thus medians were evaluated; Test type: Superiority or Other; p = 0.5811, One sample test of median (sign test)
Statistical Analysis 2: Comparison: Agalsidase Beta; Baseline versus Month 4: Analysis was performed using one sample test of median (sign test). The percent change and absolute change from baseline in urine GL-3 levels were not normally distributed and thus medians were evaluated; Test type: Superiority or Other; p = 0.7744, One sample test of median (sign test)
Statistical Analysis 3: Comparison: Agalsidase Beta; Baseline versus Month 6: Analysis was performed using one sample test of median (sign test). The percent change and absolute change from baseline in urine GL-3 levels were not normally distributed and thus medians were evaluated; Test type: Superiority or Other; p = 0.3877, One sample test of median (sign test)

4. Secondary Outcome: Percent Change From Baseline in Gastrointestinal (GI) Symptoms (Abdominal Pain, Abdominal Distention, and Bowel Irregularities) at Month 2, 4, and 6
Description: Gastrointestinal symptoms (abdominal pain, abdominal distention, and irregular bowel movements) were to be assessed by a modified version of the Irritable Bowel Syndrome (IBS) Severity Scoring System. The modified IBS Severity Scoring System is a 7-item questionnaire. The severity score calculated by summing the scores of 5 of the 7 questions. Each of the 5 questions were scored on a scale of 0 to 100, leading to a total possible score range of 0 to 500, where higher scores indicate more severe gastrointestinal symptoms. The data for this outcome measure was exploratory and to be collected in individual participant listing only.
Time Frame: Baseline, Month 2, 4, 6
Population: The data for this outcome measure was exploratory and to be collected in individual participant listing only. Analysis of this data was planned only if baseline data was collected on a large number of enrolled participants. This was not the case and therefore interpretation of these results were not possible.
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (Month 6) or early withdrawal
Description: All enrolled participants were included in the analysis.
Groups:
- Agalsidase Beta: Commercially available agalsidase beta 1.0 mg/kg administered as an intravenous infusion every 2 weeks up to Month 6.
Arm/Group | Agalsidase Beta
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Agalsidase Beta (N=15)
Infusion-associated reactions (General disorders) | 1

LIMITATIONS AND CAVEATS:
This is considered to be an exploratory study for the following reasons: it was based on a small number of participants and has been designed as an open-label, single-arm study as opposed to a two-arm crossover design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.